CLINICAL TRIAL: NCT03050801
Title: Functional Connectivity as a Biomarker of rTMS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 170055; 17-N-0055
Record Dates: First submitted 2017-02-10; First posted 2017-02-13 (Actual); Results first posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2020-06

CONDITIONS: Traumatic Brain Injury
Keywords: Explicit Memory; Implicit Memory; Memory Disorder
MeSH Terms: conditions — Brain Injuries, Traumatic; Memory Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Parietal Cortex rTMS stimulation - 1 day (Experimental): Experiment 1
  Interventions: Device: rTMS
- Parietal Cortex rTMS stimulation - 3 days (Experimental): Experiment 1
  Interventions: Device: rTMS
- Parietal Cortex rTMS stimulation - 4 days (Experimental): Experiment 1
  Interventions: Device: rTMS
- Experiment 2 - Parietal Cortex rTMS stimulation - 3 days (Experimental): Experiment 2
  Interventions: Device: rTMS
- Experiment 2 - Vertex rTMS stimulation - 3 days (Experimental): Experiment 2
  Interventions: Device: rTMS
- Experiment 2 - Prefrontal Cortex rTMS stimulation - 3 days (Experimental): Experiment 2
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — Altering the connectivity of trans-synaptic pathways

SUMMARY:
Background:

Traumatic brain injury (TBI) damages the connections between brain cells. This can lead to problems like memory loss. Repetitive transcranial magnetic stimulation (rTMS) can help improve connections between brain areas in healthy people. Researchers want to see if it can be useful in patients with memory problems after TBI.

Objective:

To see how repetitive transcranial magnetic stimulation can be used to improve the connections between parts of the brain and whether this will lead to changes in memory.

Eligibility:

Adults 18-50 years old with TBI who can speak and write in English.

Healthy volunteers the same age and English ability.

Design:

Participants will be screened with a neurological exam and may have a urine pregnancy test.

Participants with TBI will have 7-15 visits. Healthy volunteers will have 2-8 visits.

At the visits, participants will have all or some of the following:

* MRI for about 1 hour. Participants will lie in a machine that takes pictures in a magnetic field. Participants will do some memory tasks.
* Memory and attention tasks with pictures and with a computer
* Questions about their mental state and well-being
* TMS: A wire coil is held on the scalp and a short electrical current passes through it. Participants will hear a click and feel a pulling or twitch. They may be asked to make simple movements. rTMS is repeated magnetic pulses in short bursts. They will have this for about 20 minutes.

A week after the last visit, some participants will return for a memory test.

DETAILED DESCRIPTION:
Objective: To use resting state functional connectivity (FC) as a biomarker of synaptic modulation by repetitive transcranial magnetic stimulation (rTMS) in paradigms intended to improve memory and learning. Ancillary outcomes include the effects of rTMS on the interaction between the explicit implicit memory systems.

Study population: Healthy adult volunteers

Design: The study contains two experiments. Experiment 1 is designed to establish the number of rTMS sessions required to produce a meaningful change in resting parieto-hippocampal FC in healthy subjects. Experiment 2 will replicate a prior experiment which used rTMS to enhance the explicit memory system in healthy subjects, and look for potential effects on the implicit system. This intervention will be contrasted with a negative control condition (vertex stimulation) in a between-groups design.

Outcome measures: The primary outcome measure is the change in FC produced by serially applied rTMS and improvement in explicit memory. We will explore whether enhancement of the explicit system has effects on resting state connectivity in the implicit system and whether white matter integrity predicts changes in FC in healthy subjects.

ELIGIBILITY:
INCLUSION CRITERIA:

Experiments 1 and 2:

Healthy individuals

Age 18-50 (inclusive)

English speaking and writing

Experiment 3:

Age 18-50 (inclusive)

English speaking and writing

History of mild to moderate TBI

Performance 1 standard deviation below age-adjusted population norms on the

CVLT-2 within the past year from the date of visit.

EXCLUSION CRITERIA:

Any current major neurological or psychiatric disorder such as (but not limited to) stroke, Parkinson disease, Alzheimer disease, schizophrenia or major depression

History of seizure

Medications acting on the central nervous system

Ferromagnetic metal in the cranial cavity or eye, implanted neural stimulator, cochlear implant, or ocular foreign body

Implanted cardiac pacemaker or auto-defibrillator or pump

Non-removable body piercing

Claustrophobia

Inability to lie supine for 1 hour

Pregnancy, nursing, or plans to become pregnant during the study.

Members of the NINDS Behavioral Neurology Unit (BNU)

For Experiment 2: Participation in Experiment 1

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Wassermann, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Wang JX, Rogers LM, Gross EZ, Ryals AJ, Dokucu ME, Brandstatt KL, Hermiller MS, Voss JL. Targeted enhancement of cortical-hippocampal brain networks and associative memory. Science. 2014 Aug 29;345(6200):1054-7. doi: 10.1126/science.1252900. PMID 25170153
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2017-N-0055.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy Volunteers with an age range of 18-50 years were recruited for participation in Experiment 1 and 2. HV participants self-referred either directly or via the NIH Clinical Research Volunteer Program. Interested participants were pre-screened over the telephone.
  Participants with Traumatic Brain Injury were not recruited for this study, as Experiment 3 was not performed.
Pre-assignment Details: Participants were pre-screened by telephone and scheduled for consent and formal screening. Participants meeting eligibility were enrolled in the experiment. Study participants were either enrolled in Experiment 1 or 2. Experiment 1 was designed to determine the optimal number of rTMS sessions to produce a meaningful change in brain connectivity. Experiment 2 used the optimal number of rTMS sessions identified in Experiment 1, to stimulate different brain regions to study the effect on memory.
Groups:
- Experiment 1: Parietal Cortex rTMS Stimulation - 1 Day: Experiment 1
  rTMS: Altering the connectivity of trans-synaptic pathways with rTMS applied to the Parietal Cortex over 1 day
- Experiment 1: Parietal Cortex rTMS Stimulation - 3 Days: Experiment 1
  rTMS: Altering the connectivity of trans-synaptic pathways with rTMS applied to the Parietal Cortex over 3 days
- Experiment 1: Parietal Cortex rTMS Stimulation - 4 Days: Experiment 1
  rTMS: Altering the connectivity of trans-synaptic pathways with rTMS applied to the Parietal Cortex over 4 days
- Experiment 2: Parietal Cortex rTMS Stimulation - 3 Days: Experiment 2
  rTMS: Altering the connectivity of trans-synaptic pathways with rTMS applied to the Parietal Cortex over 3 days
- Experiment 2: Vertex rTMS Stimulation - 3 Days: Experiment 2
  rTMS: Altering the connectivity of trans-synaptic pathways with rTMS applied to the Vertex, over 3 days
- Experiment 2: Prefrontal Cortex Stimulation: Experiment 2
  rTMS: Altering the connectivity of trans-synaptic pathways with rTMS applied to the Prefrontal Cortex, over 3 days
Period: Experiment 1
Arm/Group | Experiment 1: Parietal Cortex rTMS Stimulation - 1 Day | Experiment 1: Parietal Cortex rTMS Stimulation - 3 Days | Experiment 1: Parietal Cortex rTMS Stimulation - 4 Days | Experiment 2: Parietal Cortex rTMS Stimulation - 3 Days | Experiment 2: Vertex rTMS Stimulation - 3 Days | Experiment 2: Prefrontal Cortex Stimulation
Started | 3 | 13 | 8 | 0 | 0 | 0
Completed | 3 | 6 | 6 | 0 | 0 | 0
Not Completed | 0 | 7 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Change of experimental design | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Unable to obtain critical rTMS measure | 0 | 0 | 2 | 0 | 0 | 0
Period: Experiment 2
Arm/Group | Experiment 1: Parietal Cortex rTMS Stimulation - 1 Day | Experiment 1: Parietal Cortex rTMS Stimulation - 3 Days | Experiment 1: Parietal Cortex rTMS Stimulation - 4 Days | Experiment 2: Parietal Cortex rTMS Stimulation - 3 Days | Experiment 2: Vertex rTMS Stimulation - 3 Days | Experiment 2: Prefrontal Cortex Stimulation
Started | 0 | 0 | 0 | 21 | 19 | 4 (Experiment 2 (Prefrontal Cortex Stimulation) was terminated early due to adverse events (intolerance of stimulation) in 2 of 4 participants.)
Completed | 0 | 0 | 0 | 15 | 15 | 2
Not Completed | 0 | 0 | 0 | 6 | 4 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Poor data quality | 0 | 0 | 0 | 4 | 1 | 0
Not completed — Discomfort during stimulation | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Experiment 2: Prefrontal rTMS Stimulation - 3 Days: Experiment 2
  rTMS: Altering the connectivity of trans-synaptic pathways with rTMS applied to the Prefrontal Cortex over 3 days
- Total: Total of all reporting groups
Arm/Group | Experiment 1: Parietal Cortex rTMS Stimulation - 1 Day | Experiment 1: Parietal Cortex rTMS Stimulation - 3 Days | Experiment 1: Parietal Cortex rTMS Stimulation - 4 Days | Experiment 2: Parietal Cortex rTMS Stimulation - 3 Days | Experiment 2: Vertex rTMS Stimulation - 3 Days | Experiment 2: Prefrontal rTMS Stimulation - 3 Days | Total
Number analyzed (Participants) | 3 | 6 | 6 | 15 | 15 | 2 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 6 | 15 | 15 | 2 | 47
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.33 (9.24) | 23.83 (2.64) | 26.67 (3.14) | 25.60 (5.46) | 24.93 (4.40) | 21.00 (2.82) | 25.27 (4.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3 | 6 | 6 | 1 | 19
  Male | 3 | 3 | 3 | 9 | 9 | 1 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 6 | 2 | 0 | 9
  Not Hispanic or Latino | 3 | 5 | 6 | 9 | 13 | 2 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 5 | 2 | 1 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 1 | 1 | 0 | 5
  White | 2 | 3 | 3 | 5 | 10 | 1 | 24
  More than one race | 0 | 0 | 1 | 1 | 2 | 0 | 4
  Unknown or Not Reported | 0 | 1 | 0 | 3 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Functional Connectivity (FC) Changes Between the Left Hippocampus and Left Parietal Cortex
Description: Transcranial Magnetic Stimulation (TMS) is a non-invasive technique which applies magnetic pulses to the brain via a coil inducing an electrical current in the brain. Stimulation is typically applied at sufficient intensity to trigger action potentials in nearby neurons.The motor threshold is defined as the minimum percentage of the stimulator output to elicit a motor evoked potential. Repetitive TMS (rTMS) was delivered at 100% of the motor evoked potential threshold with repeated magnetic pulses at a frequency of 20 Hz. Functional MRI (fMRI) measures the change in oxygenated blood in the brain; at rest these levels fluctuate over time. These fluctuations can be similar between different parts of the brain. FC is the similarity in fluctuations of these fMRI signals and suggest how strongly two regions communicate with each other. We measured how TMS can change FC between specific areas of the brain. A positive score suggests a stronger communication between regions of the brain.
Time Frame: Changes are calculated before and the day after rTMS
Population: Healthy volunteers participants
Measure: Mean (Standard Deviation); unit: Change in z-transformed R-value
Groups:
- Experiment 2: Prefrontal Cortex rTMS Stimulation - 3 Days: Experiment 2
  rTMS: Altering the connectivity of trans-synaptic pathways with rTMS applied to the Prefrontal Cortex, over 3 days
Arm/Group | Experiment 1: Parietal Cortex rTMS Stimulation - 1 Day | Experiment 1: Parietal Cortex rTMS Stimulation - 3 Days | Experiment 1: Parietal Cortex rTMS Stimulation - 4 Days | Experiment 2: Parietal Cortex rTMS Stimulation - 3 Days | Experiment 2: Vertex rTMS Stimulation - 3 Days | Experiment 2: Prefrontal Cortex rTMS Stimulation - 3 Days
Number analyzed (Participants) | 3 | 6 | 6 | 15 | 15 | 2
Change in z-transformed R-value | -0.03 (0.089) | 0.13 (0.202) | 0.02 (0.123) | -0.01 (0.109) | -0.05 (0.141) | 0.03 (0.088)

2. Primary Outcome: Associative Memory Test Score Changes
Description: Participants studied 20 face-word pairs, and after a short delay, were required to recall the word associated with each pair. The number of correctly remembered pairs was recorded. rTMS was administered over different regions of the brain over 3 days. The Associative Memory test was administered at baseline (within a week before the first rTMS session), 1 day after the last rTMS session, and again 7-14 days after the last rTMS session. We calculated improvements on this task by subtracting the number of successfully remembered pairs 1 day after stimulation from the number remembered at baseline ("Changes one day after rTMS"). We also calculated whether these improvements lasted longer by subtracting the number of successfully remembered pairs 7-14 days after stimulation from the number remembered at baseline ("Changes 7-14 days after rTMS"). Positive scores represent increases in associative memory.
Time Frame: Changes are calculated before and the day after rTMS and before and 7-14 days after rTMS
Population: Experiment 1 identified the optimal number of rTMS sessions to be applied in Experiment 2. The optimal number of rTMS sessions, i.e., 3 days, was applied to different regions of the brain in Experiment 2. Therefore, only the Experiment 2 data is reported for this outcome measure.
Measure: Mean (Standard Deviation); unit: Change in proportion of remembered pairs
Arm/Group | Experiment 2: Parietal Cortex rTMS Stimulation - 3 Days | Experiment 2: Vertex rTMS Stimulation - 3 Days | Experiment 2: Prefrontal Cortex rTMS Stimulation - 3 Days
Number analyzed (Participants) | 15 | 15 | 2
Change in proportion of remembered pairs
  Changes one day after rTMS | 0.08 (0.133) | 0.01 (0.166) | 0.03 (0.035)
  Changes 7-14 days after rTMS | 0.08 (0.173) | 0.02 (0.149) | 0.13 (0.071)

3. Secondary Outcome: Implicit Weather Prediction Task (WPT)
Description: Participants learn implicit, probabilistic relationships between stimuli and responses through feedback. 1, 2 and 3 card combinations of 4 possible cards are presented on a computer; the subject is asked to predict whether it will be rainy or fine. After each prediction, the subject receives corrective feedback. Each card is independently associated with one outcome with a fixed probability.The WPT was administered at baseline and 1 day after and 7-14 days after the last rTMS session. Scores at each time point represent the proportion of responses associated with a reward (optimal responses). We calculated improvement by subtracting the number of optimal responses 1 day after stimulation from the number at baseline (Changes one day after rTMS). We also calculated if these improvements lasted longer by subtracting the number of optimal responses 7-14 days after stimulation from the number at baseline (Changes 7-14 days after rTMS).Positive scores represent increases in implicit memory.
Time Frame: Changes are calculated before and the day after rTMS, and before and 7-14 days after rTMS
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Change in proportion of optimal response
Arm/Group | Experiment 2: Parietal Cortex rTMS Stimulation - 3 Days | Experiment 2: Vertex rTMS Stimulation - 3 Days | Experiment 2: Prefrontal Cortex rTMS Stimulation - 3 Days
Number analyzed (Participants) | 15 | 15 | 2
Change in proportion of optimal response
  Changes one day after rTMS | -0.03 (0.158) | 0.06 (0.196) | 0.06 (0.02)
  Changes 7-14 days after rTMS | -0.02 (0.143) | 0.02 (0.156) | 0.01 (0.03)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during and immediately after study procedures. Participants experiencing adverse events at completion of study procedures, were followed until AE resolution.
Arm/Group | Experiment 1: Parietal Cortex rTMS Stimulation - 1 Day | Experiment 1: Parietal Cortex rTMS Stimulation - 3 Days | Experiment 1: Parietal Cortex rTMS Stimulation - 4 Days | Experiment 2: Parietal Cortex rTMS Stimulation - 3 Days | Experiment 2: Vertex rTMS Stimulation - 3 Days | Experiment 2: Prefrontal Cortex rTMS Stimulation - 3 Days
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/13 | 0/8 | 0/21 | 0/19 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/13 | 0/8 | 0/21 | 0/19 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/13 | 0/8 | 1/21 | 0/19 | 2/4
OTHER ADVERSE EVENTS (reported when occurring in more than 4.4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experiment 1: Parietal Cortex rTMS Stimulation - 1 Day (N=3) | Experiment 1: Parietal Cortex rTMS Stimulation - 3 Days (N=13) | Experiment 1: Parietal Cortex rTMS Stimulation - 4 Days (N=8) | Experiment 2: Parietal Cortex rTMS Stimulation - 3 Days (N=21) | Experiment 2: Vertex rTMS Stimulation - 3 Days (N=19) | Experiment 2: Prefrontal Cortex rTMS Stimulation - 3 Days (N=4)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intolerance to stimulation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT03050801/Prot_SAP_000.pdf